CLINICAL TRIAL: NCT06588868
Title: Systemic Therapies in the Treatment of Cutaneous T-cell Lymphoma: an Observational Retrospective Multicenter Study
Brief Title: Systemic Therapies in the Treatment of Cutaneous T-cell Lymphoma
Acronym: FIL_CTCL
Status: Recruiting | Type: Observational
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: FIL_CTCL
Record Dates: First submitted 2024-09-03; First posted 2024-09-19 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Cutaneous T Cell Lymphoma; Cutaneous T-Cell Lymphoma/Mycosis Fungoides; Cutaneous T-Cell Lymphoma/Sezary Syndrome
Keywords: Cutaneous T Cell Lymphoma; Mycosis Fungoides; Sézary Syndrome; Retrospective; Systemic therapy; Real world
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients enrolled: Patients affected by Cutaneous T-cell Lymphoma who have received first dose of a systemic therapy, lasted at least 3 months, between 1 January 2016 and 31 December 2021 in a real life setting.

SUMMARY:
The study is designed to describe the different approaches of systemic therapies for the treatment of Cutaneous T-cell Lymphoma in real world setting.

DETAILED DESCRIPTION:
The treatment of Mycosis Fungoides (MF)/Sézary Syndrome (SS) is based on a multimodal approach through the involvement of different specialists including hematologists, dermatologists, and radiation therapists. The approach to the treatment combines different skin directed and systemic therapies (such as chemotherapies, immunomodulating agents, immunotherapies).

Although there are several well recognized therapies for the treatment of MF/SS, curative therapies are still needed. In this scenario, effective treatments that provide long term responses and disease control are still lacking. Also, International guidelines (EORTC 2017, ESMO 2018, BAD2018, NCCN) report treatment options for the different stages without recommendations of any order due to lack of evidence from clinical trials.

This study is designed to analyze the different approaches of systemic therapies for the treatment of Cutaneous T-cell Lymphoma in real world setting.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of CTCL according to the EORTC 2017 update criteria1.
* Age ≥18 years.
* Have received first dose of a systemic therapy, lasted at least 3 months, between 1 January 2016 and 31 December 2023.
* Availability of complete medical records in order to provide protocol required variables
* Signed written informed consent.

Exclusion Criteria:

* Patients not meeting the above-mentioned inclusion criteria.
* Refuse to sign a written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by Cutaneous T-cell Lymphoma who have received first dose of a systemic therapy, lasted at least 3 months, between 1 January 2016 and 31 December 2021 in real life settings
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-02-27 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
To evaluate the different systemic treatment approaches in real life settings in patients with CTCL. | The endpoint will be evaluated from the beginning to the end of the study (up to 18 months)
  Type of systemic therapies used in real-life settings for the treatment of CTCL according to disease stage.
To evaluate the different systemic treatment approaches in real life settings in patients with CTCL. | The endpoint will be evaluated from the beginning to the end of the study (up to 18 months)
  Frequency of systemic therapies used in real-life settings for the treatment of CTCL according to disease stage.
To evaluate the different systemic treatment approaches in real life settings in patients with CTCL. | The endpoint will be evaluated from the beginning to the end of the study (up to 18 months)
  Evaluation of which systemic therapies are used as first-line compared to which are used as further lines of treatment

SECONDARY OUTCOMES:
To identify real life patients' baseline clinical characteristics (e.g. CTCL subtype, cutaneous, lymphatic and blood involvement (TNMB), staging). | The endpoint will be evaluated from the beginning to the end of the study (up to 18 months)
  Frequency of baseline characteristics.
Evaluate the effectiveness of each different systemic treatment trough evaluation of best ORR attained at any time (ORRb). | The endpoint will be evaluated from the beginning to the end of the study (up to 18 months)
  Estimation of best ORR attained at any time (ORRb) of each line of systemic treatment. Kaplan-Meier estimations of time to next treatment (TTNT) and Progression free survival (PFS) according to each systemic treatment.
Overall Survival of enrolled patients. | The endpoint will be evaluated from the beginning to the end of the study (up to 18 months)
  Overall Survival
Evaluate the safety of each different systemic treatments. | The endpoint will be evaluated from the beginning to the end of the study (up to 18 months)
  Frequency of adverse events collected with the clinical course.
Impact of new drugs (brentuximab vedotin and mogamulizumab). | The endpoint will be evaluated from the beginning to the end of the study (up to 18 months)
  Estimation of best ORR attained at any time (ORRb) of each line of systemic treatment. Kaplan-Meier estimations of time to next treatment (TTNT) and Progression free survival (PFS) according to each systemic treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Pietro Quaglino, MD, Principal Investigator — SC Dermatologia U - A.O.U. Città della Salute e della Scienza di Torino
Locations (18):
- Italy (18):
  - AOU Ospedali Riuniti delle Marche - Clinica di Ematologia, Ancona
  - IRCCS Istituto Tumori Giovanni Paolo II - U.O.C. Ematologia, Bari
  - U.O.C. Dermatologia e Venereologia Universitaria - A.O.U. Policlinico Consorziale, Bari
  - Policlinico S.Orsola-Malpighi - Istituto di Ematologia, Bologna
  - ASST Spedali Civili di Brescia - S.C. Ematologia, Brescia
  - A.O. Brotzu Ospedale Businco - S.C. Ematologia e CTMO, Cagliari
  - A.O.U. Policlinico S. Marco - U.O.C. di Ematologia, Catania
  - Unità funzionale di Ematologia - Azienda Ospedaliera Universitaria Careggi, Florence
  - S.C. Dermatologia - E.O. Galliera, Genova
  - Oncoematologia - ASST Fatebenefratelli - Sacco, Milan
  - U.O.C. Dermatologia - Ospedale Maggiore Policlinico Fondazione IRCCS Ca' Granda, Milan
  - U.O.C. Clinica Dermatologica - A.O.U. di Padova, Padua
  - U.O.C Ematologia 1 - IRCCS Fondazione Policlinico San Matteo, Pavia
  - IRCCS I.F.O. San Gallicano - UOSD Porfirie e Malattie Rare, Roma
  - Skin Cancer Center - IRCCS Istituto Dermopatico dell'Immacolata, Roma
  - U.O.C. Dermatologia - A.O.U. Senese, Siena
  - A.O.U. Città della Salute e della Scienza di Torino - S.C. Dermatologia U, Torino
  - A.O.U.I. di Verona - U.O.C. Ematologia, Verona

IPD SHARING:
Plan to Share IPD: Undecided